CLINICAL TRIAL: NCT04441788
Title: A Double-Blind, Placebo-Controlled, Phase 2a Study to Assess the Safety, Tolerability, and Efficacy of ION-827359 in Patients With Mild to Moderate COPD With Chronic Bronchitis
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of ION-827359 in Participants With Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD) With Chronic Bronchitis (CB)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision to Terminate Study
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION-827359-CS2; 2020-000210-15 (EudraCT Number)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Chronic Bronchitis; Chronic Obstructive Pulmonary Disease
Keywords: Chronic Bronchitis; IONIS-ENaCRx
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Single-dose of placebo was administered by oral inhalation via nebulizer, once every week for up to 13 weeks.
  Interventions: Drug: Placebo
- ION-827359 37.5 milligrams (mg) (Experimental): Single-dose of ION-827359 37.5 mg was administered by oral inhalation via nebulizer, once every week for up to 13 weeks.
  Interventions: Drug: ION-827359
- ION-827359 75 mg (Experimental): Single-dose of ION-827359 75 mg was administered by oral inhalation via nebulizer, once every week for up to 13 weeks.
  Interventions: Drug: ION-827359

INTERVENTIONS:
Drug: ION-827359 — ION-827359 administered by oral inhalation
  Arms: ION-827359 37.5 milligrams (mg)
Drug: Placebo — Placebo administered by oral inhalation
  Arms: Placebo
Drug: ION-827359 — ION-827359 administered by oral inhalation
  Arms: ION-827359 75 mg

SUMMARY:
The purpose of this study was to evaluate the effect of ION-827359 on forced expiratory volume in 1 second (FEV1) in participants with mild to moderate COPD with CB.

DETAILED DESCRIPTION:
This was a multi-center, double-blind, placebo-controlled, randomized, Phase 2a study of ION-827359 in up to 180 participants. The participants were randomized to receive oral inhalation of either ION-827359 or placebo for up to 13 weeks. At the end of 13 weeks, participants entered a 10-week post-treatment evaluation period.

ELIGIBILITY:
Inclusion Criteria

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements
2. Males or females. Aged 40-70 inclusive at the time of informed consent
3. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or postmenopausal
4. BMI < 35.0 kg/m^2
5. Participants with a diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)

   1. Ability to perform acceptable and reproducible spirometry
   2. Post-bronchodilator (4 puffs of albuterol) spirometry at Screening demonstrating the following:

   i. FEV1/ forced vital capacity (FVC) ratio of < 0.70 ii. FEV1 ≥ 50% and ≤ 90% of predicted normal
6. Clinically stable COPD in the 4 weeks prior to Screening (Visit 1)
7. Current and former smokers with smoking history of ≥ 20 pack years
8. Meet SGRQ definition of CB
9. CAT score ≥ 10

Exclusion Criteria

1. Clinically significant abnormalities in medical history (e.g., previous acute coronary syndrome within 6 months of screening, congestive heart failure, major surgery within 3 months of Screening) or physical examination
2. Screening laboratory results as follows, or any other clinically significant abnormalities in screening laboratory values that would render a subject unsuitable for inclusion

   1. Urine protein/creatinine (P/C) ratio ≥ 0.3 mg/mg. In the event of P/C ratio above this threshold eligibility may be confirmed by a quantitative total urine protein measurement of < 300 mg/24 hr
   2. Positive test (including trace) for blood on urinalysis. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
   3. alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, alkaline phosphatase (ALP), serum creatinine, blood urea nitrogen (BUN) > 1.5 × upper limit of normal (ULN)
   4. Platelet count < LLN
   5. Serum potassium > 5.2 mmol/L
   6. Estimated GFR < 60 mL/min (as determined by the Cockcroft-Gault Equation for creatinine clearance)
   7. A positive PCR test for SARS-CoV-2 at any time prior to randomization
3. Any active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to first day Study Drug product is administered to the participant (Study Day 1)
4. Unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator
5. Clinically important pulmonary disease other than COPD
6. Asthma as a primary or main diagnosis according to the Global Initiative for Asthma (GINA) guidelines (GINA 2011) or other accepted guidelines. Participants with a past medical history of asthma (e.g. childhood or adolescence) may be included
7. Treatment with systemic corticosteroids and/or antibiotics, and/or hospitalization for a COPD exacerbation within 4 weeks prior to enrolment (Visit 1)
8. Acute upper or lower respiratory infection requiring antibiotics or antiviral medication within 4 weeks prior to enrolment (Visit 1)
9. Long term oxygen therapy (LTOT)
10. Participants participating in, or scheduled for, an intensive (active) COPD rehabilitation program (participants who are in the maintenance phase of a rehabilitation program are eligible to take part)
11. Concomitant medication restrictions: Oral anticoagulants, oral steroids (e.g. prednisone or Medrol), theophylline, chronic azithromycin, or roflumilast
12. Have any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the Study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Czechia (5):
  - MediTrial s.r.o., Jindřichův Hradec
  - Plicni ambulance Kralupy, Kralupy nad Vltavou
  - CEFISPIRO s.r.o., Lovosice
  - Plicni Ambulance Rokycany, s.r.o., Rokycany
  - PNEUMOLOGIE VARNSDORF s.r.o., Varnsdorf
- Germany (7):
  - Pneumologisches Studienzentrum Markgrafenstrasse, Berlin
  - MECS Research GmbH, Berlin
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Hamburger Institut far Therapieforschung GmbH, Hamburg
  - KLB Gesundheitsforschung Lubeck GmbH, Lübeck
  - IKF Pneumologie Mainz Helix Medical Excellence Center Mainz, Mainz
  - ZMS-Zentrum fur medizinische Studien GmbH, Warendorf
- Hungary (2):
  - Csongrad Megyei Mellkasi Betegsegek Szakkorhaza, Deszk
  - Selye Janos Korhaz, Rendelointezet, Komárom
- Queen Anne Street Medical Centre, Heart Lung Center, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 participants were randomized at 11 study centers in Czech Republic, Germany, Hungary and the United Kingdom.
Pre-assignment Details: Of the 60 randomized participants, one was randomized but did not receive study treatment as the participant was ineligible. The study included a 2-week screening period (including a diet-stabilization period), a 12-week treatment period, and a 10-week post-treatment evaluation period.
Period: Overall Study
Arm/Group | Placebo | ION-827359 37.5 Milligrams (mg) | ION-827359 75 mg
Started | 20 | 21 | 19
Completed | 3 | 4 | 3
Not Completed | 17 | 17 | 16
Not completed — Voluntary Withdrawl | 0 | 1 | 0
Not completed — Ineligibility | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Study Terminated by Sponsor | 16 | 16 | 12

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who were randomized and received at least 1 dose of study drug.
Groups:
- ION-827359 37.5 mg: Single-dose of ION-827359 37.5 mg was administered by oral inhalation via nebulizer, once every week for up to 13 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg | Total
Number analyzed (Participants) | 19 | 21 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (4.54) | 61.8 (5.86) | 61.8 (5.39) | 61.6 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 5 | 21
  Male | 10 | 14 | 14 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 21 | 19 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 19 | 21 | 18 | 58
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] — FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
  liters | 1.8317 (0.4670) | 1.9311 (0.6608) | 1.6536 (0.3498) | 1.8097 (0.5193)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Primary Time Point in Forced Expiratory Volume in 1 Second (FEV1) Compared to Placebo
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Baseline was defined as the last non-missing measurement prior to the first study drug administration. The primary time point was defined as the average of weeks 13 and 14. FAS=Full analysis set.
Time Frame: From Baseline up to average of Weeks 13 and 14
Population: FAS=all randomized participants who had ≥1 dose of study drug(ION 827359/placebo),≥1 post-Baseline efficacy assessment(i.e.,post-Baseline FEV1,Exacerbations of Chronic pulmonary Disease Tool[EXACT]Respiratory Symptoms[E-RS]score,Chronic Obstructive Pulmonary Disease[COPD]Assessment Test[CAT]score,or St.George's Respiratory Questionnaire-COPD Specific[SGRQ-C score],post-bronchodilator FEV1).Overall number analyzed:number of participants with data available for analyses in this outcome measure.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 5 | 5 | 4
liters | 0.0642 (0.2506) | -0.0240 (0.3581) | 0.1336 (0.1087)

2. Secondary Outcome: Change From Baseline in the Exacerbations of Chronic Pulmonary Disease Tool (EXACT) Respiratory Symptoms (E-RS) Daily Symptom Diary Total Score to the Primary Time Point
Description: The E-RS scale is a participant-reported outcome (PRO) designed to measure the symptoms of participants with chronic obstructive pulmonary disease (COPD). The E-RS utilizes 11 respiratory symptom items from the existing and validated 14-item EXACT, which measures symptoms of exacerbation. The E-RS total score quantifies respiratory symptom severity, and 3 domains assess breathlessness (comprised of 5 items, score range [0-17]), cough and sputum (comprised of 3 items, score range [0-11]), and chest symptoms (comprised of 3 items, score range [0-12]). The E-RS was collected on the daily e-diary. The total score was derived by summing the 11-item scores and ranged between 0 to 40 with higher values indicating severe respiratory symptoms. The primary time point was defined as the average of weeks 13 and 14.
Time Frame: From Baseline up to average of weeks 13 and 14
Population: FAS included all randomized participants who received at least 1 dose of study drug (ION-827359 or placebo) and who had at least 1 post-Baseline efficacy assessment (i.e., post-Baseline FEV1 assessment, E-RS score, CAT score, or SGRQ-C score). Overall number of participants analyzed is the number of participants with data available for analyses in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 4 | 5 | 4
score on a scale | -1.08 (1.171) | -1.41 (2.486) | -1.99 (4.217)

3. Secondary Outcome: Change From Baseline in the Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) to the Week 14 Time Point
Description: The CAT is an eight-item questionnaire that was completed by the participant and is designed to quantify the impact of COPD symptoms on the health status of participants. Each item is rated on a 6-point scale ranging from 0 (no impairment) to 5 (maximum impairment). The total CAT score is calculated by summing the scores of all items and ranges from 0 to 40. Higher scores indicate a severe condition (more severe impact of COPD on a participant's life).
Time Frame: From Baseline to Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 5 | 5 | 3
score on a scale | -2.6 (2.51) | -0.6 (3.78) | 0.0 (1.73)

4. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire - COPD Specific (SGRQ-C) Total Score to the Week 14 Time Point
Description: The SGRQ is a participant completed, a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in participants with obstructive airway disease. The shorter 40-item version (SGRQ-C) which does not specify a Recall Period and has been validated specifically for COPD participants was used in this study. It consists of 40 items each weighted from 0 to a possible maximum of 100. Items 1-7 produced the symptoms score, 9-12 the activity score, and items 8, 10, 11, 13 and 14 the impacts score. Each component sub-score was calculated as a percentage of the summed weights of each item out of the sum of the maximum possible weight for that component (range 0-100). The total score was calculated by summing the weights to all positive responses in each component, where a positive item indicated the presence of symptoms, expressed as a percentage (range 0-100). Higher scores indicated a worse outcome (more limitations)
Time Frame: From Baseline to Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 5 | 5 | 3
score on a scale | -15.93 (19.515) | -1.74 (3.839) | -0.76 (2.350)

5. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV1
Description: Post-bronchodilator FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation after administration of bronchodilator. Baseline was defined as the last non-missing measurement prior to the first study drug administration.
Time Frame: From Baseline to end of treatment (EOT) [Up to Week 14]
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 3 | 5 | 3
liters | 0.0663 (0.0685) | 0.0320 (0.2379) | 0.1180 (0.1006)

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for ION-827359
Time Frame: Days 1 and 85
Population: Pharmacokinetic (PK) population included all participants who were randomized and received at least 1 dose of active study drug (ION-827359) and had at least 1 evaluable PK sample collected and analyzed with reportable result. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 6 | 6
nanogram per milliliter (ng/mL)
  Day 1 | 85.6 (198) | 203 (52.6)
  Day 85: number analyzed (Participants) | 1 | 2
  Day 85 | 53.5 (NA) — The geometric coefficient of variation was not estimable due to lower number of participants. | 195 (124)

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration for ION-827359
Time Frame: Days 1 and 85
Population: PK population included all participants who were randomized and received at least 1 dose of active study drug (ION-827359) and had at least 1 evaluable PK sample collected and analyzed with reportable result. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Median (Full Range); unit: hours
Arm/Group | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 6 | 6
hours
  Day 1 | 1.54 [0.567 to 2.05] | 1.64 [0.667 to 2.12]
  Day 85: number analyzed (Participants) | 1 | 2
  Day 85 | 1.98 [1.98 to 1.98] | 3.11 [1.73 to 4.48]

8. Secondary Outcome: AUC[0-24h]: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours for ION-827359
Time Frame: Days 1 and 85
Population: PK population consisted of all the participants who were randomized and received at least 1 dose of active study drug (ION-827359) and had at least 1 evaluable PK sample collected and analyzed with reportable result. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 6 | 6
hours*nanogram per milliliter (h*ng/mL)
  Day 1 | 528 (190) | 1323 (66.0)
  Day 85: number analyzed (Participants) | 1 | 2
  Day 85 | 312 (NA) — The geometric coefficient of variation was not estimable due to lower number of participants. | 2416 (252)

9. Secondary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) Based on Severity
Description: An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of medicinal (investigational) product, whether or not the AE is considered related to the medicinal (investigational) product. A TEAE is defined as any AE starting or getting worse on or after the first dose of the study drug. The severity of a TEAE was assessed by the investigator and classified into one of the following: mild, moderate, and severe.
Time Frame: Up to Week 24
Population: Safety population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 19 | 21 | 19
percentage of participants
  Mild | 10.5 | 14.3 | 15.8
  Moderate | 52.6 | 38.1 | 63.2
  Severe | 10.5 | 0 | 5.3

10. Secondary Outcome: Percentage of Participants With Clinically Significant Change in Laboratory Values
Description: Laboratory parameters for serum chemistry, hematology, urinalysis, coagulation, complement, and lipids were assessed.
Time Frame: Up to Week 24
Population: Safety population included all participants who are were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 19 | 21 | 19
percentage of participants | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Clinically Significant Change in Vital Sign Parameters
Description: Vital signs included assessment of heart rate, blood pressure, respiratory rate, and temperature.
Time Frame: Up to Week 24
Population: Safety population included all participants who are were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 19 | 21 | 19
percentage of participants | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings
Description: ECG parameters of ventricular rate, PR interval, QRS duration, QT, or QTc were assessed.
Time Frame: Up to Week 24
Population: Safety population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
Number analyzed (Participants) | 19 | 21 | 19
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: Safety population included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Placebo | ION-827359 37.5 mg | ION-827359 75 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/21 | 1/19
Other Adverse Events (participants affected / at risk) | 14/19 | 8/21 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | ION-827359 37.5 mg (N=21) | ION-827359 75 mg (N=19)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | ION-827359 37.5 mg (N=21) | ION-827359 75 mg (N=19)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Burning sensation (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Cyst (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 1
FEV1/FVC ratio decreased (Investigations) | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Vaccination complication (Immune system disorders) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Product taste abnormal (Product Issues) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated based on the toxicology findings from a 9-month study and participants who had not completed the treatment period were instructed to terminate dosing and return for an end of study visit, followed by the 10-week follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT04441788/Prot_SAP_000.pdf